CLINICAL TRIAL: NCT00335101
Title: Renal Effects of Three Iodinated Contrast Media (CM) in Patients at Risk Undergoing Coronary Angiography
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor Decision to withdraw study (comparative product withdrawn from the market)
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: GE-012-091
Record Dates: First submitted 2006-06-06; First posted 2006-06-08 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease (CAD); Renal Impairment; Diabetes Mellitus
Keywords: Coronary Artery Disease (CAD), Renal Impairment, Serum creatinine (SCr), Iodixanol, Ioversol, Iopromide, Contrast Induced Nephropathy (CIN)
MeSH Terms: conditions — Coronary Artery Disease; Renal Insufficiency; Diabetes Mellitus | interventions — iodixanol; ioversol; iopromide

INTERVENTIONS:
Drug: Iodixanol, Ioversol, Iopromide

SUMMARY:
The study is to evaluate and compare the effects on kidney function of three iodinated contrast media (CM) in patients at risk of kidney damage evaluating serum creatinine (Scr) concentrations up to three days after CM administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a combination of DM (type I or II) and renal impairment (RI), defined as SCr ≥150 µmol/L (1.7 mg/dL) for men and ≥133 µmol/L (1.5 mg/dL) for women or creatinine clearance (CrCl) ≤50 mL/min calculated according to Cockroft-Gault formula, referred for coronary angiography with or without PCI.

Exclusion Criteria:

* Concurrent administration of potentially nephroprotective or nephrotoxic drugs is not allowed. Subjects undergoing dialysis or kidney transplantation or with CrCl < 20 mL/min will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06

PRIMARY OUTCOMES:
Primary endpoint:
Maximum peak increase in SCr from baseline up to day 3.
Secondary endpoints:
Change in SCr from baseline to day 2 and to day 3
Number of subjects with contrast-induced nephropathy (CIN)
Quality of diagnostic information

SECONDARY OUTCOMES:
Coronary Artery Disease (CAD)
Renal Impairment
Diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pignot, PhD, Study Director — GE Healthcare; Johnny Gibbs, Jr., CCRA, Study Director — GE Healthcare
Locations (2):
- GE Healthcare, Princeton, New Jersey, United States
- GE Healthcare, Munich, Germany